CLINICAL TRIAL: NCT06834646
Title: Comparison of 30-day Morbidity and Mortality in Cancer Patients Based on Emergency Department Location: Referring Oncology Hospital vs Other Hospitals.
Brief Title: Comparison of 30-day Morbidity and Mortality in Cancer Patients Based on Emergency Department Location
Acronym: COVER
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240971; IDRCB: 2024-A01679-38 (Other: ANSM)
Record Dates: First submitted 2025-02-05; First posted 2025-02-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cancer Remission
Keywords: Emergency Department; Cancer; Mortality; morbidity and mortality in Cancer
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who visit the ED of the refereing oncologic hospital
- Patients who visit another ED

SUMMARY:
Patients being followed for cancer account for 2.8% of emergency admissions in France. An acute episode that triggers a visit to the emergency department may be related to the progression of the disease, or to complications of treatment. The management of these patients is often complex and requires a degree of expertise. Emergency departments specialising in the management of cancer complications have been set up, and now deal exclusively with patients treated at their centres. However, for geographical or logistical reasons, patients with cancer are likely to consult a non-specialist emergency department and/or one located outside the cancer care centre. In this case, the emergency doctor may not have access to the oncology file, and care in the emergency department and downstream services may be sub-optimal. Studies have shown a positive impact on the quality of care and prognosis of patients thanks to the cancer centre's expertise. However, the effect of the centre on a cancer patient who visits the emergency department has never been studied. This is particularly true if the emergency department where the patient is seen is located in the cancer follow-up centre.

The primary objective of the COVER study is to investigate the impact of the location of the emergency department where the patient is seen for their prognosis.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 or over admitted to an emergency department with cancer that has been active or in remission for less than a year.

Exclusion Criteria:

- Opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for cancer and consulting the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of days alive spent outside the hospital | 1 month

SECONDARY OUTCOMES:
Occurrence of a new/ unscheduled consultation | 30 days
Length of hospitalisation | 90 day
Unscheduled consultation or hospitalization emergency department discharge | 7 days
Unexpected death | 7 days
Secondary admission to the intensive care unit during the initial hospitalization following the emergency visit | 7 days
Occurence of organ failure | 7 days
Quality of life with QLQ-C30 | 90 days
  QLQ-C30
Mortality | 30 days
Mortality | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpêtrière Emergency department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided